CLINICAL TRIAL: NCT05694000
Title: Deep Brain Stimulation of the Ventral Hippocampus in Treatment-resistant Schizophrenia: Exploring the Glutamatergic/GABAergic Mechanisms
Brief Title: Hippocampus DBS in Treatment-resistant Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Dengtang LIU, Chief Psychiatrist and Professor, Shanghai Mental Health Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 82171496
Record Dates: First submitted 2022-12-09; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Treatment-resistant Schizophrenia
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- On-Stimulation (Active Comparator): Disease condition is assessed with stimulation turned "on".
  Interventions: Device: On-Stimulation
- Off-Stimulation (Placebo Comparator): Disease condition is assessed with stimulation turned "off".
  Interventions: Device: Off-Stimulation

INTERVENTIONS:
Device: On-Stimulation — The surgical electrode implanted in hippocampus by a pulse generating device is "on".
  Arms: On-Stimulation
Device: Off-Stimulation — The surgical electrode implanted in hippocampus by a pulse generating device is "off".
  Arms: Off-Stimulation

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of hippocampus-targeted deep brain stimulation (DBS) in treatment-resistant schizophrenia. The main question it aims to answer are:

* whether patients with treatment-resistant schizophrenia can benefit from hippocampus-targeted DBS;
* what is the neural and electrophysiological mechanism underlying the treatment effect of hippocampus-targeted DBS.

DETAILED DESCRIPTION:
The first phase of the study will consist of DBS surgery. Participants will receive electrodes implantation in bilateral ventral hippocampus. Continuous stimulation will be applied to optimize and individualize the stimulus parameters. This period is anticipated between 3 and 6 months.

The next phase will consist of the crossover study. Patients who respond to DBS will be randomly assigned to two groups, for a period of 3 months: on stimulation group and off stimulation group. Patients will then be crossed over to the other group for a further 3 months.

Participants will receive PET-CT, clinical assessment and cognitive tests at the main study points to evaluate treatment efficacy and patient tolerance, and to reveal the underlying mechanism of the treatment effect of DBS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 55 years.
* Having a diagnosis of schizophrenia according to DSM-IV criteria
* Having a chronic, recurrent course of disease with a five-year minimum duration
* Determined to be treatment-resistant as demonstrated by:

  1. Persistence of positive symptoms which have not responded to appropriate treatments for at least 2 years.
  2. Inadequate response from adequate trials of two different classes of antipsychotic drugs (not including clozapine), at least 8 weeks.
  3. Inadequate response from adequate trial of clozapine, at least 3 months, or unable to tolerate clozapine because of intolerable side effects.
  4. Presence of persistent positive symptom defined as i) requiring a score of 4 (moderate) or more on at least 2 of the next PANSS items: delusions, conceptual disorganization, hallucinatory behavior, suspiciousness and unusual thought content; or as ii) requiring a score of 6 (severe) or more on at least 1 of the above PANSS items.
* Maintaining stable pharmacological treatment for two months preceding screening visit.
* Informed consent

Exclusion Criteria:

* Neurological disease
* Severe physical illness
* Contraindications to neurosurgery, MRI or PET-CT;
* Substance abuse or dependence
* Mental retardation
* Female patients who are pregnant or breastfeeding
* Severe suicide risk and tendencies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Scale to assess changes in clinical symptoms; response to DBS is defined as a 20% reduction from baseline in PANSS score

SECONDARY OUTCOMES:
Clinical Global Impression-Schizophrenia (CGI-SCH) Scale | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Scale to assess changes in symptoms' severity, global improvement or change
Clinician-Rated Dimensions of Psychosis Symptom severity (CRDPS) Scale | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Scale to assess different dimensions and severity of symptoms
The Chinese version of Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Battery of neuropsychological tests to assess changes in cognition
Cerebral metabolism(PET-CT scans) | Baseline, 24 weeks, 48 weeks
  Assessment of changes in metabolic levels of glutamate, GABA and dopamine in the whole brain using PET-CT

OTHER OUTCOMES:
Adverse events (AEs) | Baseline, 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Any unexpected medical problem that may happen during DBS treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dengtang Liu, Principal Investigator — liudengtang@smhc.org.cn
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Lu C, Zhai Z, Zhuo K, Xiang Q, Xue J, Zhao Y, Lang L, Shao C, Chen L, Liu D. Deep brain stimulation of Hippocampus in Treatment-resistant Schizophrenia (DBS-HITS): protocol for a crossover randomized controlled trial. BMC Psychiatry. 2024 Nov 25;24(1):847. doi: 10.1186/s12888-024-06318-6. PMID 39587538